CLINICAL TRIAL: NCT02302170
Title: A Phase Ⅲ Clinical Trial for Efficacy, Immunogenicity, Safety and Immune Persistence of Oral Recombinant Helicobacter Pylori Vaccine in Chinese Children Aged From 6-15 Years Old.
Brief Title: A Phase Ⅲ Clinical Trial With Oral Recombinant Helicobacter Pylori Vaccine in Chinese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: National Institutes for Food and Drug Control, China (Other); Kangwei Biological Technology (Other); Third Military Medical University (Other)
Responsible Party: Principal Investigator, Fengcai Zhu, Vice director of Jiangsu Province Centers for Disease Control and Prevention, Jiangsu Province Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TMMUHP03
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: H. Pylori Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- H. pylori vaccine in children (Experimental): H. pylori vaccine (15mg/dose) in children between 6-15 years of age
  Interventions: Biological: H. pylori vaccine
- placebo in children (Placebo Comparator): placebo (0mg/dose) in children between 6-15 years of age
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: H. pylori vaccine
  Other Names: Oral Recombinant Helicobacter Pylori Vaccine
  Arms: H. pylori vaccine in children
Biological: placebo
  Arms: placebo in children

SUMMARY:
Helicobacter pylori (H. pylori) is a Gram-negative, microaerophilic bacterium that persistently colonizes the human stomach; more than half the human population is infected worldwide. H. pylori infection is a risk factor for the development of gastritis, peptic ulcer, gastric mucosa-associated lymphoid tissue lymphoma, and gastric cancer.

The phaseⅠand Ⅱclinical trial of oral recombinant Helicobacter pylori vaccine had completed in Jiangsu Province in China. The data from phaseⅠand Ⅱclinical trial suggested that the oral recombinant Helicobacter pylori vaccine had a clinically acceptable safety and good immunogenicity for health adults and children. To further explore the safety and immunogenicity profile of this vaccine, a phase Ⅲ clinical trial was conducted.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a Gram-negative, microaerophilic bacterium that persistently colonizes the human stomach; more than half the human population is infected worldwide. H. pylori infection is the major risk factor for the development of gastritis, peptic ulcer, gastric mucosa-associated lymphoid tissue lymphoma, and gastric cancer.

At present, the main clinical treatment for H. pylori infection is the application of antibiotics and bismuth agent or H+ antagonists. Due to the widespread drug resistance, toxic side effects, high medical costs as well as poor patient compliance, it is unworkable to practice antibiotics therapy for H. pylori eradication on every patient. Vaccination is the most effective way for prevention H. pylori infection.

Since H. pylori were found, great attention has been given to the H. pylori vaccine, scientists worldwide have made great efforts to develop both prophylactic and therapeutic H. pylori vaccine. Numerous H. pylori vaccine approaches have been studied, including inactivated whole cell H. pylori vaccine, genetic engineering subunit vaccine, live vector vaccines. Urease is considered to be an excellent candidate antigen for vaccine against H. pylori. However, no vaccine against H. pylori has been used in clinic.

The phaseⅠand Ⅱclinical trial of oral recombinant Helicobacter pylori vaccine had completed in Jiangsu Province in China. The data from phaseⅠand Ⅱclinical trial suggested that the oral recombinant Helicobacter pylori vaccine had a clinically acceptable safety and good immunogenicity for children. To further explore the safety and immunogenicity profile of this vaccine, a phase Ⅲ clinical trial was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged from 6-15 years old as established by medical history and clinical examination
* The subjects' guardians are able to understand and sign the informed consent
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting before vaccination

Exclusion Criteria:

Exclusion criteria for the first dose

* Subject who has a medical history of stomach illness
* Positive in either serology ELISA test for Helicobacter pylori diagnose kit or 13C urea breath test
* Subject who has suffered from heart, liver, and kidney disease
* Subject who has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine (for example: mannitol)
* Subject who is suffering from thrombocytopenia or other coagulation disorder
* Subject who has a diminished function of the immune system or autoimmune disease
* Subject who is suffering from congenital deformities, developmental disorders or serious chronic diseases
* Family history of seizures or progressive neurological disease
* Severe malnutrition or dysgenopathy, major congenital defects or serious chronic illness, including perinatal brain damage
* Any acute infections in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 month
* Any prior administration of other research medicines in last 1 month
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Exclusion criteria for the second and third dose Subjects will not be eligible for the second or third dose if any of following happened after first dose

* Subject who had allergic reaction to the last dose
* Any situation meet the exclusion criteria occurred after the last dose
* Subject who had any serious adverse events related to the vaccination
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4464 (Actual)
Dates: Start 2004-12; Primary Completion 2006-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The occurrence of Helicobacter pylori infection in participants one year after three-dose vaccinations. | one year after the third dose

SECONDARY OUTCOMES:
The immune response of anti-UreB IgG antibodies in serum after three-dose vaccinations in the immunogenicity subset of participants | 1 month after the third dose
  seroconversion rates, GMTs, GMFI of anti-UreB IgG antibodies in serum after three-dose vaccinations in the immunogenicity subset of participants at month 1.
The immune response of anti-UreB sIgA antibodies in saliva after three-dose vaccinations in the immunogenicity subset of participants | 1 month after the third dose
  conversion rates, GMTs, GMFI of anti-UreB sIgA antibodies in saliva after three-dose vaccinations in the immunogenicity subset of participants at month 1
The immune response of anti-UreB IgG antibodies in serum three-dose vaccinations in the immunogenicity subset of participants. | 6 months after the third dose
  seroconversion rates, GMTs, GMFI of anti-UreB IgG antibodies in serum after three-dose vaccinations in the immunogenicity subset of participants at month 6
The immune response of anti-UreB IgA antibodies in saliva after three-dose vaccinations in the immunogenicity subset of participants | 6 months after the third dose
  To evaluate conversion rates, GMTs, GMFI of anti-UreB sIgA antibodies in saliva after three-dose vaccinations in the immunogenicity subset of participants at month 6
The immune response of anti-UreB IgG antibodies in serum after three-dose vaccinations in the immunogenicity subset of participants | 12 months after the third dose
  seroconversion rates, GMTs, GMFI of anti-UreB IgG antibodies in serum after three-dose vaccinations in the immunogenicity subset of participants at month 12
The immune response of anti-UreB sIgA antibodies in saliva after three-dose vaccinations in the immunogenicity subset of participants | 12 months after the third dose
  conversion rates, GMTs, GMFI of anti-UreB sIgA antibodies in saliva after three-dose vaccinations in the immunogenicity subset of participants at month 12
Frequency of adverse reactions after taking the H. pylori vaccines in children | within 3 days after each vaccination
  Frequency of adverse reactions within 3 days after taking the H. pylori vaccines in children
Occurrence of serious adverse reactions after taking the H. pylori vaccines in children | From day 0 to One year after the third dose
  Occurrence of serious adverse reactions within one year after the third dose in children
Anti-UreB IgG antibodies persistency in serum after three-dose vaccinations in the immunogenicity subset of participants | 24 months after the third dose
  seroconversion rates, GMTs, GMFI of anti-UreB IgG antibodies in serum after three-dose vaccinations in the immunogenicity subset of participants at month 24
Anti-UreB IgA antibodies persistency in saliva after three-dose vaccinations in the immunogenicity subset of participants | 24 months after the third dose
  conversion rates, GMTs, GMFI of anti-UreB sIgA antibodies in saliva after three-dose vaccinations in the immunogenicity subset of participants at month 24
Anti-UreB IgG antibodies persistency in serum after three-dose vaccinations in the immunogenicity subset of participants | 36 months after the third dose
  seroconversion rates, GMTs, GMFI of anti-UreB IgG antibodies in serum after three-dose vaccinations in the immunogenicity subset of participants at month 36
Anti-UreB IgA antibodies persistency in saliva after three-dose vaccinations in the immunogenicity subset of participants | 36 months after the third dose
  To evaluate conversion rates, GMTs, GMFI of anti-UreB sIgA antibodies in saliva after three-dose vaccinations in the immunogenicity subset of participants at month 36
The occurrence of Helicobacter pylori infection in participants in the second year after three-dose vaccinations. | in the second year after the third dose
The occurrence of Helicobacter pylori infection in participants in the third year after three-dose vaccinations. | in the third year after the third dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zeng M, Mao XH, Li JX, Tong WD, Wang B, Zhang YJ, Guo G, Zhao ZJ, Li L, Wu DL, Lu DS, Tan ZM, Liang HY, Wu C, Li DH, Luo P, Zeng H, Zhang WJ, Zhang JY, Guo BT, Zhu FC, Zou QM. Efficacy, safety, and immunogenicity of an oral recombinant Helicobacter pylori vaccine in children in China: a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2015 Oct 10;386(10002):1457-64. doi: 10.1016/S0140-6736(15)60310-5. Epub 2015 Jun 30. PMID 26142048